CLINICAL TRIAL: NCT01490879
Title: A Randomized, Prospective, Double-blind, Vehicle-controlled, Dose-ranging, Multi-center Study to Assess the Safety and Clinical Effect of Nexagon® in the Treatment of Subjects With a Diabetic Foot Ulcer
Brief Title: A Study to Investigate the Safety and Clinical Effect of Nexagon® as a Topical Treatment for Subjects With a Diabetic Foot Ulcer (DUNE)
Acronym: DUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OcuNexus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEX-ULC-011
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Foot Ulcers
Keywords: DFU; Diabetic Foot Ulcer; Ulcers; Foot Ulcers; chronic wound; wounds; Nexagon; CoDa
MeSH Terms: conditions — Diabetic Foot; Ulcer; Foot Ulcer; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nexagon® Low Dose (Experimental): Twice weekly applications of Nexagon® low dose in addition to off-loading using a Removable Cast Walker
  Interventions: Drug: Nexagon® Low Dose
- Nexagon® Medium Dose (Experimental): Twice weekly applications of Nexagon® medium dose in addition to off-loading using a Removable Cast Walker
  Interventions: Drug: Nexagon® Medium Dose
- Nexagon® High Dose (Experimental): Twice weekly applications of Nexagon® high dose in addition to off-loading using a Removable Cast Walker
  Interventions: Drug: Nexagon® High Dose
- Nexagon® vehicle (Placebo Comparator): Twice weekly applications of Nexagon® vehicle in addition to off-loading using a Removable Cast Walker
  Interventions: Drug: Nexagon® vehicle

INTERVENTIONS:
Drug: Nexagon® Low Dose — Twice weekly, topical application of Nexagon® low dose in addition to a Removable Cast Walker
  Arms: Nexagon® Low Dose
Drug: Nexagon® Medium Dose — Twice weekly, topical application of Nexagon® medium dose in addition to a Removable Cast Walker
  Arms: Nexagon® Medium Dose
Drug: Nexagon® High Dose — Twice weekly, topical application of Nexagon® high dose in addition to a Removable Cast Walker
  Arms: Nexagon® High Dose
Drug: Nexagon® vehicle — Twice weekly, topical application of Nexagon® vehicle in addition to a Removable Cast Walker
  Arms: Nexagon® vehicle

SUMMARY:
This study is for Type I or Type II diabetic subjects with with a diabetic foot ulcer. The study is being done to determine if Nexagon® plus standard of care is more effective than placebo plus standard of care. Standard of care will include debridement of the ulcer, standardized dressings and standardized off-loading using a Removable Cast Walker.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diabetes mellitus (Type I or II)
2. HbA1c of less than or equal to 12.0%
3. Diagnosis of neuropathic foot ulcer with partial or complete neuropathy
4. Cutaneous ulcer on the plantar or dorsal aspect of the foot or toe that is greater or equal to 1.0cm2 and less than or equal to 8.0 cm2 in area at the end of the screening period and is full thickness with no exposed ligament, tendon, joint capsule or bone. Surface area will be measured by digital planimetry.
5. The Medical Monitor(or delegate)must confirm that the reference diabetic foot ulcer (RDFU)is suitable for inclusion after reviewing digital photographs
6. Wound bed consisting of completely viable tissue or one where completely viable tissue will be achieved by the end of the screening period.
7. An Ankle Branchial Index (ABI) of greater or equal to 0.80 in concert with a bi- or tri-phasic Doppler flow pattern; or adequate circulation as demonstrated by any of the following methods: peri-wound transcutaneous partial pressure oxygen (TcpO2)greater or equal to 40 mmHg; or a toe pressure of greater or equal to 40 mmHg; or skin perfusion pressure of greater or equal to 40 mmHg.
8. Ulcer present for 4 weeks or more or less than or equal to 12 months.
9. Willing to wear a Removable Cast Walker (RCW) between study visits for the duration of the study.
10. Signed informed consent form.

Exclusion Criteria:

1. Any unstable medical condition that would cause the study to be detrimental to the subject.
2. Decrease in RDFU size by more than 40% or increase in the ulcer size by more than 40% during the 14-day screening period as measured by digital planimetry.
3. Ulcers caused primarily by untreated vascular insufficiency or ulcers with an etiology not related to diabetes.4. Ulcers above the ankle.

5. Ulcers that cannot be effectively off-loaded using the cast walker and sole insert provided in this study (ulcers not located on the weight bearing surface of the foot do not require off-loading).

6. Ulcers on the toes not accessible for photography (e.g. in the web space). 7. Presence of other ulcers within 2cm of the perimeter of the RDFU. 8. BMI > 45 9. Cannot tolerate or will not comply with the off-loading method, or non-compliance with standard or care.

10.The RDFU is infected (clinical assessment of infection)and/or biopsy proof of greater than 100,000 organisms per gram of tissue during the screening period.

11. Subjects presenting with the clinical characteristics of cellulitis at the ulcer site. 12. Necrosis, purulence, or sinus tracts that cannot be removed by debridement.13. Definite or suspected osteomyelitis within any wound located anywhere on the subjects body.14. Acute Charcot's neuroarthropathy as determined by clinical and/or previous radiographic examination.

15. Severe Charcot deformity or rocker bottom foot with an associated plantar mid-foot or heel ulcer.

16. Revascularization surgery on the leg with the wound to be treated less than or equal to 4 weeks prior to the start of the screening period.

17. Requirement for concurrent topical antimicrobials to treat the RDFU after the end of the screening period.

18. Received dermal substitute or living skin equivalent (e.g. Dermagraft® or Apligraf®) within 14 days prior of the start of the screening period.

19. Severe complications of diabetes that in the opinion of the Investigator could interfere with wound healing or impede the subject's participation.

20. Subjects on concurrent immunosuppressive therapy to include oral corticosteroid therapy equivalent to greater than 5 mg/day of prednisone.

21. Any history of radiation therapy to the foot. 22. Female subjects who are pregnant or lactating. 23. Pre-menopausal women not using effective birth control methods as determined by the Investigator. 24. Life expectancy of < 12 months. 25. Subjects on renal replacement therapy. 26. Cancer within the last 3 years except basal and squamous cell carcinoma. 27. Cancer within the RDFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Reference Diabetic Foot Ulcer (RDFU) complete closure determined by Investigator Assessment | Within 12 weeks

SECONDARY OUTCOMES:
Percentage change in RDFU surface area | Within 12 weeks
Time to RDFU complete closure | Within 12 weeks
Percentage of granulation tissue in RDFU | 12 weeks
Incidence of ulcer recurrence | 12 weeks post-closure
Incidence of adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM MD PhD, Principal Investigator — S.A.L.S.A. , University of Arizona, Tucson, AZ
Locations (25):
- United States (9):
  - Associated Foot and Ankle Specialists, LLC, Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - Center For Clinical Research Inc., Castro Valley, California
  - Advanced Foot Care and Clinical Research Center, Fresno, California
  - Barry University Clinical Research, Hialeah, Florida
  - Univeristy of Miami, Miller School of Medicine, Dermatology Research, Miami, Florida
  - Doctors Research Network, South Miami, Florida
  - Advanced Foot and Ankle Center, Las Vegas, Nevada
  - Houston Foot and Ankle Care, Houston, Texas
- Russia (9):
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - City Clinical Hospital #13, Moscow
  - Endocrinology Science Center, Moscow
  - Endocrinology Clinic of Moscow, Department of Healthcare, Moscow
  - Moscow Medical University n.a., Moscow
  - Federal bureau of medical and social expertise, Moscow, Moscow
  - St Petersburg City Hospital of St Elizabeth, Saint Petersburg
  - St Petersburg Diagnostic Center, Saint Petersburg
  - Voronezh Regional Clinical Consultative Diagnostic Center, Voronezh
- Ukraine (7):
  - Cherkasy Regional Clinical Hospital, Endocrinology Department, Cherkasy
  - Dnipropetrovsk Regional Clinical Hospitaln. a. I.I. Mechnikov, Dnipropetrovsk
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Regional Clinical Hospital, Cardiovascular Surgery Department, Kharkiv
  - Kyiv City Clinical Hospital #1, Kyiv
  - Institute of Endocrinology and Methabolism n.a. V.P. Komisarenko, Clinical Diabetology Department, Kyiv
  - Zaporizhzhya City Clinical Hospital #9, Zaporizhzhya